CLINICAL TRIAL: NCT00482066
Title: A Pilot Study Examining the Effect of Abatacept in ANCA Associated Vasculitis
Brief Title: Abatacept in ANCA Associated Vasculitis
Acronym: ABAVAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funders withdrew funding due to slow recruitment
Sponsor: Imperial College London (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: cro632; 2006-001859-35 (EudraCT Number); BMS protocol No: IST110 (Other Grant/Funding Number: Bristol Myers Squib funder)
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-03

CONDITIONS: ANCA-associated Vasculitis
Keywords: Wegener's granulomatosis; Microscopic polyangiitis; Churg Strauss Syndrome; ANCA
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Abatacept (Orencia)
  Interventions: Drug: Abatacept (Orencia)
- 2 (Placebo Comparator): saline placebo
  Interventions: Drug: Abatacept (Orencia)

INTERVENTIONS:
Drug: Abatacept (Orencia) — 500mg for patients under 60kg 750mg for patients 60-100kg
  1g for patients>100kg given as i.v. infusion over 30 minutes at day 0, 14, 28 and then monthly for a further 11 months 914 infusions in total) placebo groups receive saline only I.v.

SUMMARY:
The purpose of this study is to investigate whether abatacept can prevent relapse in patients with ANCA associated vasculitis(AAV). This is a randomised double blinded placebo controlled trial.

DETAILED DESCRIPTION:
The drugs that are normally used to treat patients with AAV are quite effective, but up to 20% of patients relapse within 18 months. The drugs used can also have significant side effects. Abatacept, also known as CTLA4Ig, acts by blocking vital costimulatory signals required for T lymphocytes to be activated. As ANCA associated vasculitis is believed to be an autoimmune condition and dependent on autoreactive T cells, there is some reason to believe this drug would be effective. Abatacept has already received a license by the FDA for use in Rheumatoid arthritis where it has proven to be effective even in patients unresponsive to Etanercept (TNF blockade).

120 patients with AAV will be invited to take part in this study, from hospitals in the UK and Europe. The patients will receive standard therapy with methotrexate and steroids as well as 12 months of abatacept or placebo. They will be followed for a further 12 months.

The primary objective of this study is to assess the relapse rate over 24 months, in patients with acute AAV, presenting at first diagnosis or relapse, in the two arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute AAV, presenting at first diagnosis or relapse, defined by clinical presentation
* ANCA positivity (anti-MPO or anti-PR3 positive)
* BVAS score of > 8.

Exclusion Criteria:

* Severe life-threatening disease, i.e. lung haemorrhage at the time of presentation, renal impairment with SCr>150 micromol/l, or severe CNS dysfunction thought to be due to vasculitis.
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological or cerebral disease, or other medical conditions that might place the subject at unacceptable risk for participation in this study.
* Any other non-vasculitic multisystem autoimmune disease
* Serious acute or bacterial infection unless treated and completely resolved with antibiotics prior to enrolment
* With any severe chronic or recurrent bacterial infection
* With Hepatitis B or C or HIV
* With Herpes zoster infection that resolved less than 2 months prior to enrolment
* Subjects who have received any live vaccines within 3 months of the first dose of study medication or who will have need of a live vaccine at any time in the year following enrolment
* Subjects with current clinical or laboratory evidence of active or latent tuberculosis (TB) and subjects with a history of active TB treated within the last 3 years
* With any previous malignancy, with the exception of non-melanoma skin malignancies, adequately treated previously
* Subjects with a mammogram that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded following additional evaluations. Mammograms (females only) must be performed within 6 months of study entry or if documentation is not on file.
* With MTX treatment in prior 3 months
* Subjects with prior therapy with rituximab, anti-TNF therapy, or IL-1 receptor antagonists within last year or cyclophosphamide within last six months
* Subjects with a history of intolerance to methotrexate
* Subjects who have at any time received treatment with abatacept
* Subjects who have received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose
* Subject receiving approved or investigational biologics
* Subjects with any of the following laboratory values:

  * Hgb < 8.5 g/dL.
  * WBC < 3,000/mm3 (3 x 109/L)
  * Platelets < 100,000/mm3 (100 x 109/L).
  * Serum ALT or AST > 2 times upper limit of normal.
  * Any other laboratory test results that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study.
* Subjects participating concurrently in another clinical trial
* Pregnancy, breast feeding or inadequate contraception if female.
* Allergy to a study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Relapse rate over 24 months. | 2 years

SECONDARY OUTCOMES:
Proportion of patients in sustained remission (i.e. remission at 3 months sustained for 6 months and remission at 6 months sustained for a further 12 months); | 2 years
Time to remission; | 2 years
The average steroid dosage at 6 months, 1 year, 18 months and 2 years in abatacept and placebo groups respectively; | 2 years
Time to ANCA negativity by immunofluorescence or negative anti-PR3 or anti-MPO Ab test by ELISA. | 2 years
Proportion of patients defaulting to cyclophosphamide (MMF, azathioprine or other rescue) therapy. | 2 years
Proportion of patients unable to stick with trial protocol. | 2 years
Degree of chronic disease activity | 2 years
Health related quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan Salama, Study Director — Imperial College London
Locations (1):
- Imperial College London, Hammersmith Hospital, London, United Kingdom